CLINICAL TRIAL: NCT00072072
Title: A Phase I Trial Of A COX-2 Inhibitor (Celecoxib) In Combination With An EGFR Inhibitor (OSI-774) In Metastatic Non-Small Cell Lung Cancer
Brief Title: Celecoxib and Erlotinib in Treating Patients With Stage IIIB or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000335434; UCLA-0306083
Record Dates: First submitted 2003-11-04; First posted 2003-11-06 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2006-01

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Celecoxib; Erlotinib Hydrochloride

INTERVENTIONS:
Drug: celecoxib
Drug: erlotinib hydrochloride

SUMMARY:
RATIONALE: Celecoxib may stop the growth of cancer by stopping blood flow to the tumor. Erlotinib and celecoxib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Combining celecoxib with erlotinib may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of celecoxib when given together with erlotinib in treating patients with stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the biologically active dose of celecoxib administered with erlotinib in patients with stage IIIB or IV non-small cell lung cancer.
* Determine the toxicity profile of this regimen in these patients.

Secondary

* Determine the clinical activity of this regimen, in terms of reduction in tumor burden, in these patients.
* Correlate biological endpoints with cyclooxygenase-2 and epidermal growth factor receptor inhibition in patients treated with this regimen.

OUTLINE: This is a nonrandomized, dose-escalation study of celecoxib.

Patients receive oral erlotinib once daily and oral celecoxib twice daily on days 1-28. Treatment repeats every 4 weeks for 2 courses in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease may continue treatment beyond 2 courses at the investigator's discretion.

Cohorts of 3-6 patients receive escalating doses of celecoxib until the maximum tolerated dose (MTD) and biologically active dose (BAD) are determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity (DLT). The BAD is defined as the maximum decrease in the level of PGE_2 where no DLT occurs.

Patients are followed every 2 months.

PROJECTED ACCRUAL: A total of 21-27 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-small cell lung cancer (NSCLC)

  * Stage IIIB or IV
* Measurable disease
* Progressive disease after at least 2 prior standard chemotherapy regimens OR refused standard chemotherapy
* No active CNS metastases

PATIENT CHARACTERISTICS:

Age

* 21 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 mg/dL
* Transaminases no greater than 2.5 times upper limit of normal (ULN)
* PT and/or PTT no greater than 1.5 times ULN

Renal

* Creatinine no greater than 2 mg/dL

Cardiovascular

* No New York Heart Association class III or IV cardiac disease
* No myocardial infarction within the past year
* No symptomatic ventricular arrhythmia
* No symptomatic conduction abnormality

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior gastrointestinal ulceration, bleeding, or perforation
* No hypersensitivity to celecoxib, sulfonamides, aspirin, other NSAIDs, or other reagents used in this study
* No concurrent disease or medical condition that would preclude study treatment or compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* More than 4 weeks since prior chemotherapy

Endocrine therapy

* More than 4 weeks since prior corticosteroids
* No concurrent steroids (including chronic use)

  * Concurrent topical steroids allowed

Radiotherapy

* More than 4 weeks since prior radiotherapy

Surgery

* Not specified

Other

* More than 4 weeks since prior non-cytotoxic investigational agents
* More than 3 days since prior nonsteroidal anti-inflammatory drugs (NSAIDs)
* No prior cyclooxygenase-2 (COX-2) inhibitors for metastatic NSCLC
* No prior epidermal growth factor receptor inhibitor for metastatic NSCLC
* No concurrent COX-2 inhibitors
* No concurrent NSAIDs
* No concurrent fluconazole or lithium

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-08; Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A. Figlin, MD, FACP, Principal Investigator — Jonsson Comprehensive Cancer Center; Karen Rickard, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States

REFERENCES:
- [Result] Reckamp KL, Krysan K, Morrow JD, Milne GL, Newman RA, Tucker C, Elashoff RM, Dubinett SM, Figlin RA. A phase I trial to determine the optimal biological dose of celecoxib when combined with erlotinib in advanced non-small cell lung cancer. Clin Cancer Res. 2006 Jun 1;12(11 Pt 1):3381-8. doi: 10.1158/1078-0432.CCR-06-0112. PMID 16740761